CLINICAL TRIAL: NCT06509412
Title: Nd:YAG Laser Versus Diode Laser Assisted New Attachment Procedure (Lanap) in the Management of Stage II Periodontitis: Randomized Controlled Clinical Trial
Brief Title: Nd:YAG Laser Versus Diode Laser Assisted New Attachment Procedure (Lanap) in the Management of Stage II Periodontitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nada Shaban (Other)
Responsible Party: Sponsor-Investigator, Nada Shaban, Master's candidate of Periodontology, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2/2023
Record Dates: First submitted 2024-07-14; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LANAP surgical protocol using ND:YAG 1064 laser (Experimental)
  Interventions: Device: LANAP surgical protocol using ND:YAG 1064 laser
- LANAP surgical protocol using diode 940 laser (Experimental)
  Interventions: Device: LANAP surgical protocol using diode 940 laser
- Scaling and root planing (Active Comparator)
  Interventions: Procedure: Scaling and root planing (SRP)

INTERVENTIONS:
Device: LANAP surgical protocol using ND:YAG 1064 laser — A free running pulsed, 1064 nm wavelength-specific ND:YAG laser (Light walker AT)* with an attached 320 µm diameter optical glass fiber attached to a metallic hand piece with a flexible tip, which will be set at 3:4 -watt average power, 20 HZ, and a 100-600 µs pulse duration
  Arms: LANAP surgical protocol using ND:YAG 1064 laser
Device: LANAP surgical protocol using diode 940 laser — Diode laser (Biolase) with 940 nm wavelength, a thin flexible fiber-optic cable 300 μm was attached with a power average set at 0.5-1 watt, in continuous mode, and 20 HZ
  Arms: LANAP surgical protocol using diode 940 laser
Procedure: Scaling and root planing (SRP) — Scaling and root planing (SRP) using ultrasonic device (Woodpecker USD-P Led Ultrasonic Scaler Ende) at moderate setting and with appropriate tips and also hand curettes will be used for root planning.
  Arms: Scaling and root planing

SUMMARY:
Aim of the study was to assess and compare the clinical and microbiological changes following Laser assisted new attachment procedure (LANAP®) using diode 940 nm versus ND:YAG 1064 nm, and to compare the outcome to conventional periodontal therapy

ELIGIBILITY:
Inclusion Criteria:

* Periodontal diagnosis of stage II periodontitis.
* Residual periodontal pocket ≥4 mm, 3-4 mm clinical attachment loss with horizontal bone loss higher than 15% in radiography.
* O'Leary plaque index <10%.

Exclusion Criteria:

* Patients with furcation involvement.
* Class II/III tooth mobility.
* Smokers who smoke more than 10 cigarettes per day.
* Patients with any systemic condition possibly affecting the outcome of periodontal therapy.
* Patients who had received any local or systemic anti-inflammatory medications or antibiotics within the last 6 months.
* Alcohol consumers.
* Pregnant or lactating women.
* Patients with parafunctional habits.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Microbiological assessment of Treponima denticola | up to six months
  Sub-gingival dental plaque biofilm will be collected using size 50 paper point after ensuring a good isolation of the operating field, and sample will be placed in sterile microcentrifuge tubes containing phosphate buffered saline to be transferred immediately to the Microbiology Laboratory of Alexandria University Hospitals. Microcentrifuge tubes will be vortexed for 5 minutes then 200 ul of resulting suspension will be subjected to DNA extraction using QIAamp DNA Minikit (Qiagen, Germany). Specific PCR primers targeting gingival plaque-associated oral microbiota (Treponima denticola Td) will be used in SYBER green real-time PCR. Amplification of the 16SrRNA gene will be used as the denominator against which the amplification of other bacteria will be estimated. The bacterial relative quantification will be calculated automatically by Rotor-gene software and expressed as relative fold difference.
Microbiological assessment of Prevotella intermedia | up to six months
  Sub-gingival dental plaque biofilm will be collected using size 50 paper point after ensuring a good isolation of the operating field, and sample will be placed in sterile microcentrifuge tubes containing phosphate buffered saline to be transferred immediately to the Microbiology Laboratory of Alexandria University Hospitals. Microcentrifuge tubes will be vortexed for 5 minutes then 200 ul of resulting suspension will be subjected to DNA extraction using QIAamp DNA Minikit (Qiagen, Germany). Specific PCR primers targeting gingival plaque-associated oral microbiota (Prevotella intermedia Pi) will be used in SYBER green real-time PCR. Amplification of the 16SrRNA gene will be used as the denominator against which the amplification of other bacteria will be estimated. The bacterial relative quantification will be calculated automatically by Rotor-gene software and expressed as relative fold difference.
Gingival health | up to six months
  The gingival index (Löe and Silness,1967) will be used to assess the degree of gingival inflammation. Each tooth is examined and scored (0-3), where 0 = normal gingiva; 1 = mild inflammation: slight change in color, slight edema, no bleeding on probing; 2 = moderate inflammation: redness, edema, and glazing, or bleeding on probing; 3 = severe inflammation: marked redness and edema, tendency toward spontaneous bleeding and ulceration
Clinical attachment loss (CAL) | up to six months
  This is assessed using a Williams probe from a fixed reference point on the crown to the base of the pocket. Pocket severity is classified by the extent of clinical attachment loss in millimeters (0= normal, 1 or 2 mm = slight, 3 or 4 mm = moderate, ≥ 5 mm = severe).
Pocket probing depth (PPD) | up to six months
  This is measured from the margin of the gingiva to the base of the pocket using a Williams probe. The normal probing sulcus depth is considered to range from 1 to 3 mm in healthy gingiva.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt